CLINICAL TRIAL: NCT04061616
Title: Transcultural Validation of the Physical Activity Scale for Individuals With Physical Disabilities (PASIPD) in French: The PASIPD-Fr
Acronym: PASIPD-Fr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PASIPD-Fr
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2019-08

CONDITIONS: Physical Disability; Neurological Diseases or Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): All the participants volunteer to participate to the study that were included.
  Interventions: Behavioral: PASIPD-Fr

INTERVENTIONS:
Behavioral: PASIPD-Fr — Fill-out the PASIPD-Fr self questionaire twice (2 completions at a 2-week interval)

SUMMARY:
The Physical Activity Scale for Individuals With Physical Disabilities (PASIPD) is a scale that has been developped and validated in English to quantify the level of physical activity for people with physical disabilities. The investigators aimed to translate and validate a French transcultural version of the PASIPD (PASIPD-Fr) through a rigourous process following international recommendations for cross-cultural translation and adaptation of questionnaires.

DETAILED DESCRIPTION:
For the translation, permission to proceed was obtained, and translation was conducted in consultation with the developers. The investigators proceed to a first translation of the initial scale from English to French with two French native bilingual physicians that resulted in a unique french translation. An English native bilingual physicians proceeded to a back translation from French to English. This version have been sent to the developers who agreed that this back translated version was faithful to the original scale.

For the validation, the investigators used the international recommendations for cross-cultural translation and adaptation of questionnaires. Population was individuals with neurological disease (stroke, multiple sclerosis, Parkinson disease and neuromuscular disorders) with significant in physical disability. Patients were invited in an ambulatory setting. Data collected for every participant included demographic and general variables (age, sex, level, cause and time since neurological disease, walking capacities and aid), scores of a physical performance tests (10 Meter Walking Test, 10 MWT) and the 4 self-administered questionnaires: the Dijon Physical Activity Scale (PAS) the Activities-specific Balance Confidence (ABC) Scale, the Medical Outcome Study Short Form 12 " (MOS SF-12) and the Hospital Anxiety and Depression (HAD) scale.

Face validity was assessed using verbal feedbacks from physician and patients, and the mean time to fill-out the scale.

Criterion validity was assessed with correlation and discrimination analysis between the scores for the PASIPD-Fr and the Dijon PAS.

Construct validity was assessed using the correlation with scores of instruments that measure various aspects related to and physical activity (convergent validity) such as the self-reported questionaires ABC, SF-12 and HAD scales and also the 10 MWT.

For consistency and reliability, the investigators calculated the Cronbach α coefficient and calculated the ICC between 2 completions at a 2-week interval.

Sample calculation was based on an expected ICC > 0.9, which required 50 participants to reject the hypothesis that the actual ICC is < 0.6, which corresponds to the lower limit for a "good" reproducibility.

ELIGIBILITY:
Inclusion Criteria:

* Patient who received research information
* Patient affiliated to a social security system
* Patient over 18 years of age
* Patients with physical disabilities (Act No. 2005-102 on equal rights and opportunities)
* Individuals with the following disease: stroke survivors, multiple sclerosis, neuromuscular disease and idiopathic Parkinson's disease

Exclusion Criteria:

* Patient not affiliated to a social security system.
* Patients under guardianship or curators or protection of justice.
* Lack of informed information about the study
* Alteration of higher functions or sensory disturbance making it impossible to understand and adhere to the research protocol
* A severe medical condition that significantly alters functional abilities (severe heart failure, respiratory failure, unstable metabolic disorders such as active renal failure) and involves a life-threatening condition in the short to medium term (progressive neoplastic pathology, unstable systemic disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Criterion validity (correlation) | Both scales (PASIPD-Fr and Dijon PAS) were filled-out in a single point of time within a period of time of 12 months (study time frame)
  The Dijon PAS assesses the level of physical activity in the general population, the elderly and is recommended after a stroke. To test the criterion validity of the PASIPD-Fr, the investigators calculated the Pearson correlation coefficient (PCC) between the scores for the PASIPD-Fr and the Dijon PAS.
Criterion validity (discrimination) | Both scales (PASIPD-Fr and Dijon PAS) were filled-out in a single point of time within a period of time of 12 months (study time frame)
  The Dijon PAS assesses the level of physical activity in the general population, the elderly and is recommended after a stroke. To test the criterion validity of the PASIPD-Fr, the investigators used the repeated measures ANOVA to check for differences between inactive, moderately active ang highly active individuals (respectively score <10, 10-20 and >20 over 30 on Dijon PAS) with Tukey post-hoc tests.
Test-retest reliability | The PASIPD-Fr was administered twice at a 2-week interval within a period of time of 12 months (study time frame)
  The investigators calculated the intraclass coefficient (ICC) between 2 completions of the PASIPD-Fr questionnaire at a 2-week interval.

SECONDARY OUTCOMES:
Construct validity 10TMWT | Both PASIPD-Fr questionaire and 10MWT test were assessed in a single point of time within a period of time of 12 months (study time frame)
  The 10 Meter Walk Test is is a performance measure used to assess walking speed in metres per second over a short distance.To test the criterion validity of the PASIPD-Fr, the investigators calculated the Pearson correlation coefficient (PCC) between the scores for the PASIPD-Fr and the 10MWT
Construct validity ABC-S | Both PASIPD-Fr questionaire and ABC-S scale were filled-out in a single point of time within a period of time of 12 months (study time frame)
  The Activities-specific balance confidence (ABC) scale is a subjective measure of confidence in performing various ambulatory activities without experiencing a sense of unsteadiness.To test the criterion validity of the PASIPD-Fr, the investigators calculated the Pearson correlation coefficient (PCC) between the scores for the PASIPD-Fr and the ABC-S
Construct validity HAD | Both PASIPD-Fr questionaire and HAD scale were filled-out in a single point of time within a period of time of 12 months (study time frame)
  The Hospital Anxiety and Depression scale (HAD) is used to determine the levels of anxiety and depression that a person is experiencing. To test the criterion validity of the PASIPD-Fr, the investigators calculated the Pearson correlation coefficient (PCC) between the scores for the PASIPD-Fr and the HAD
Construct validity MOS SF12 | Both PASIPD-Fr questionaire and MOS SF12 scale were filled-out in a single point of time within a period of time of 12 months (study time frame)
  The Medical Outcome Study Short Form 12 " (MOS SF-12) is used to measure mental and physical health. To test the criterion validity of the PASIPD-Fr, the investigators calculated the Pearson correlation coefficient (PCC) between the scores for the PASIPD-Fr and the MOS SF12
Internal consistency | The PASIPD-Fr scale was filled-out in a single point of time within a period of time of 12 months (study time frame)
  To measure the internal consistency (homogeneity) of the PASIPD-Fr, based on average inter-item correlations and the number of items.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided